CLINICAL TRIAL: NCT00284258
Title: Phase II/III Trial of CPT-11/5-FU/l-LV (FOLFIRI) Versus CPT-11/TS-1 (IRIS) as Second Line Chemotherapy of Unresectable Colorectal Cancer
Brief Title: Phase II/III Trial of CPT-11/5-FU/l-LV Versus CPT-11/TS-1 as Second Line Chemotherapy of Unresectable Colorectal Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01023010 / TOP-003
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; titanium silicide; Fluorouracil

ARMS (2):
- 1 (Experimental): CPT-11 and TS-1
  Interventions: Drug: CPT-11 and TS-1
- 2 (Active Comparator): CPT-11, 5-FU and l-LV
  Interventions: Drug: CPT-11, 5-FU and l-LV

INTERVENTIONS:
Drug: CPT-11 and TS-1 — TS-1 was administered orally at 40-60 mg twice daily for 14 days with a rest period of 14 days as one course. CPT-11 was administered intravenously 125 mg per square meter at day1 and day14 in 4 weeks as one course.
  Arms: 1
Drug: CPT-11, 5-FU and l-LV — Patients were administered FOLFIRI every 2 weeks in one course. FOLFIRI:CPT-11 150 mg per square meter on day1 with l-LV 200 mg per square meter administered as a 2-hour infusion before 5-FU 400 mg per square meter administered as an intravenous bolus injection, and 5-FU 2400 mg per square meter as a 46-hour infusion immediately after 5-FU bolus injection on day1 in 2 weeks.
  Arms: 2

SUMMARY:
This study is designed as Phase II/III. Phase II is aimed to evaluate safety and efficacy of IRIS, and feasibility of FOLFIRI. Phase III is aimed to verify inferiority of the progression free survival of IRIS in comparison with FOLFIRI.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer
* Locally advanced and/or metastatic colorectal cancer
* Have prior chemotherapy as first line treatment
* No prior irinotecan administration
* Able to take oral medication
* Age 20 to 75
* Performance status 0 or 1 (ECOG)
* WBC 3,000-12,000 / mm^3
* Platelet ≥100,000 / mm^3
* AST and ALT ≤ 100 IU/L
* Creatinine ≤ 1.2 mg/dL
* Bilirubin ≤ 1.5 mg/dL

Exclusion Criteria:

* Prior radio therapy for colorectal cancer
* Other malignancies in the past 5 years
* Serious illness or medical condition

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2006-01; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Progression free survival | every course for first three courses, then every other course

SECONDARY OUTCOMES:
Over all survival, Response rate, Adverse event, Medical economy | adverse events will be collected during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Sugihara, MD, PhD, Principal Investigator — Tokyo Medical and Dental University Hospital
Locations (1):
- Saku Central Hospital, Saku, Nagano, Japan

REFERENCES:
- [Result] Muro K, Boku N, Shimada Y, Tsuji A, Sameshima S, Baba H, Satoh T, Denda T, Ina K, Nishina T, Yamaguchi K, Takiuchi H, Esaki T, Tokunaga S, Kuwano H, Komatsu Y, Watanabe M, Hyodo I, Morita S, Sugihara K. Irinotecan plus S-1 (IRIS) versus fluorouracil and folinic acid plus irinotecan (FOLFIRI) as second-line chemotherapy for metastatic colorectal cancer: a randomised phase 2/3 non-inferiority study (FIRIS study). Lancet Oncol. 2010 Sep;11(9):853-60. doi: 10.1016/S1470-2045(10)70181-9. Epub 2010 Aug 12. PMID 20708966
- [Derived] Yasui H, Muro K, Shimada Y, Tsuji A, Sameshima S, Baba H, Satoh T, Denda T, Ina K, Nishina T, Yamaguchi K, Esaki T, Tokunaga S, Kuwano H, Boku N, Komatsu Y, Watanabe M, Hyodo I, Morita S, Sugihara K. A phase 3 non-inferiority study of 5-FU/l-leucovorin/irinotecan (FOLFIRI) versus irinotecan/S-1 (IRIS) as second-line chemotherapy for metastatic colorectal cancer: updated results of the FIRIS study. J Cancer Res Clin Oncol. 2015 Jan;141(1):153-60. doi: 10.1007/s00432-014-1783-3. Epub 2014 Aug 9. PMID 25106731